CLINICAL TRIAL: NCT05032755
Title: Using Very Low Nicotine Cigarettes to Disrupt the Pain-smoking Reinforcement Cycle
Brief Title: Low Nicotine Cigarettes, Smoking, and Chronic Pain
Acronym: VLNCPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00108705; R21DA052729 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Smoking, Cigarette
MeSH Terms: conditions — Chronic Pain; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLNC Group (Experimental): Participants in this condition will be provided with Spectrum NRC102/103 (nonmenthol/menthol) cigarettes, which have a nicotine content of approximately 0.4 mg/g tobacco with reported nicotine yield (ISO) of 0.03 +/- 0.01 mg and a tar yield of 9 +/- 1.5. Participants will be asked to smoke only study cigarettes for 4 weeks.
  Interventions: Other: SPECTRUM NRC 102/103 investigational cigarettes
- NNC Group (Active Comparator): Participants in this condition will be provided with Spectrum NRC600/601 (non-menthol/menthol) cigarettes, which have a nicotine content of approximately 15.8 mg/g tobacco with reported nicotine yield (ISO) of 0.8 +/- 0.15 mg and a tar yield of 10.5 +/- 1.5.
  Interventions: Other: SPECTRUM NRC 600/601 investigational cigarettes

INTERVENTIONS:
Other: SPECTRUM NRC 102/103 investigational cigarettes — Very low nicotine content (nonmenthol/menthol) SPECTRUM investigational cigarettes
  Arms: VLNC Group
Other: SPECTRUM NRC 600/601 investigational cigarettes — Normal nicotine content (nonmenthol/menthol) SPECTRUM investigational cigarettes
  Arms: NNC Group

SUMMARY:
The purpose of this study is to evaluate the effects of switching to very low nicotine content (VLNC) cigarettes versus normal nicotine content (NNC) cigarettes on experiences with craving, withdrawal, and pain among individuals with chronic back pain who smoke cigarettes daily.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effects of very low nicotine content (VLNC) cigarettes on the dynamic associations between smoking, pain, and withdrawal among daily smokers with chronic (> 3 months) non-cancer back pain (n=48). Participants will complete an initial screening session to determine eligibility, followed by a baseline abstinence session in which measures of pain and withdrawal will be assessed following 24 hrs abstinence from smoking. At the conclusion of this session participants will receive training in ecological momentary assessment (EMA) procedures and software will be installed on their smartphone. Participants will then complete a 1-week baseline period, in which they will complete EMA while continuing to smoke usual brand cigarettes. During EMA, participants will receive 6 randomly spaced daily prompts, with 15 questions to complete about smoking behavior, mood, and current pain. In addition, participants will be asked to use their smartphone to indicate whenever they are about to smoke a cigarette. Three of these cigarettes each day will be randomly selected for assessment: in these cases participants will be asked to respond to the same 15 question before and after smoking the cigarette. Participants will also complete end of day questionnaires.

After the 1 week baseline period, participants will be randomly assigned to four weeks of either VLNCs (n=24) or normal nicotine content (NNC) cigarettes (n=24). During this period, participants will be asked to smoke only study cigarettes. Participants will attend weekly laboratory visits to provide biochemical verification of cigarette adherence (urine samples) and complete questionnaires. Study cigarettes will also be provided and collected at these visits. Two of the four weekly urine samples will be selected for analysis. Participants will also complete EMA during weeks 1 and 4 of study cigarette use. End of day questionnaires will continue throughout the 4 weeks.

At the conclusion of the study, participants will attend a final laboratory visit after abstaining from smoking for 24 hours. During this session, self-report measures of pain, craving, and withdrawal will be assessed, along with biochemical verification (breath sample) of abstinence.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of non-cancer chronic (>3 months) back pain (confirmed in medical record or by current provider);
* Pain duration of >=3 months with an average intensity of >/= 4/10 or worst pain >/=6/10 as assessed by Graded Chronic Pain Scale (GCPS);
* smoking at least 10 cigarettes per day for > 2 years;
* expired breath CO concentration > 10 ppm;
* have an iPhone or Android smartphone capable of running EMA software

Exclusion Criteria:

* actively taking steps to quit smoking;
* inability to attend all required experimental sessions;
* report of significant health problems;
* systolic blood pressure > 160 or diastolic blood pressure > 100;
* resting heart rate > 100;
* breath alcohol level > 0.0;
* current use of opioid pain relievers;
* lifetime history of bipolar or psychotic disorder;
* current unstable psychiatric disorder as assessed by the MINI;
* use of non-cigarette tobacco products > 8 times in the past 30 days;
* current use of nicotine replacement therapy (NRT) or other smoking cessation strategy;
* use of Spectrum investigational cigarettes in the past year;
* quit attempt in the past 30 days resulting in > 3 days abstinence;
* past year alcohol or substance use disorder;
* use of illegal drugs as measured by urine drug screen;
* pain complaint due to specific medical conditions (e.g., cancer, rheumatoid arthritis, complex regional pain syndrome);
* spine surgery within the past year or planned surgery within the timeframe of the study;
* current disability litigation pending;
* positive pregnancy test among women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Sweitzer, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Duke University Medical Center and the surrounding area from August, 2023 through May, 2024.
Pre-assignment Details: A total of 40 participants were determined to be eligible and enrolled in the study. Of these, 5 withdrew prior to randomization due to scheduling difficulty (n=2), PI decision following repeated no-shows (n=1), inability to abstain from smoking for the baseline abstinent visit (n=1) and loss to contact (n=1).
Period: Overall Study
Arm/Group | VLNC Group | NNC Group
Started | 19 | 16
Completed | 19 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLNC Group | NNC Group | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (9.69) | 49.8 (8.15) | 50.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 15 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Smoked Per Day
Description: Average number of cigarettes smoked per day over the past week, as reported on timeline follow-back interview at each weekly visit
Time Frame: Weekly for 5 weeks
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
cigarettes/day
  Week 1 | 14.5 (5.54) | 17.2 (7.39)
  Week 2 | 16.4 (8.99) | 20.3 (6.49)
  Week 3 | 13.5 (7.15) | 23.4 (5.86)
  Week 4 | 13.8 (7.84) | 22.5 (5.87)
  Week 5 | 14.0 (8.95) | 23.8 (8.09)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p < .0001, Mixed Models Analysis; Model includes random intercepts; beta estimate = 1.902, Standard Error of Mean 0.398 — Estimation parameter is beta estimate for group by visit interaction term

2. Primary Outcome: Weekly Measures of Cigarette Dependence as Assessed by the Fagerstrom Test of Cigarette Dependence (FTCD)
Description: The FTCD is a widely used 6-item measure of dependence, with total scores ranging from 0 (low dependence) to 10 (high dependence)
Time Frame: Weekly for 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 | 4.95 (2.12) | 5.56 (1.59)
  Week 2 | 4.32 (2.31) | 5.88 (1.78)
  Week 3 | 4.11 (2.35) | 6.19 (1.56)
  Week 4 | 3.84 (2.34) | 6.12 (1.67)
  Week 5 | 4.16 (2.34) | 6.25 (1.73)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p < .0001, Mixed Models Analysis — Group is entered as a between-subjects factor and Visit is included as a repeated factor with 5 levels. Baseline pain and FTCD scores, assessed at screening, are included along with sex as covariates; Model includes random intercepts; beta estimate = 0.368, Standard Error of Mean 0.08 — Estimation parameter is beta estimate for group by visit interaction term

3. Primary Outcome: Weekly Ratings of Withdrawal Symptoms as Measured by the Minnesota Tobacco Withdrawal Scale
Description: The MNWS is a 7-item measure of withdrawal symptoms, with responses indicated on a likert scale ranging from 0 (none) to 4 (severe). The total score ranges from 0 to 28, with higher scores indicating greater withdrawal symptoms.
Time Frame: Weekly for 5 visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 | 12.05 (5.64) | 10.69 (4.25)
  Week 2 | 12.42 (6.31) | 10.38 (4.72)
  Week 3 | 12.32 (6.25) | 12.38 (3.95)
  Week 4 | 9.84 (6.27) | 11.25 (5.53)
  Week 5 | 10.42 (5.64) | 10.69 (3.44)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.065, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model includes random intercepts; beta estimate = 0.672, Standard Error of Mean 0.362 — Estimation parameter is beta estimate for group by visit interaction term

4. Primary Outcome: Weekly Changes in Pain Intensity as Measured by the Past-week Version of the Brief Pain Inventory (BPI)
Description: The BPI is a well-validated 11-item self-report measure. Pain intensity is calculated as the average of 3 items (worst pain, least pain, and average pain). Scores are averaged with the total score ranging from 0 to 10 with higher scores indicating more pain.
Time Frame: Weekly for 5 visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 | 5.1 (1.89) | 4.04 (1.02)
  Week 2 | 4.97 (1.8) | 3.88 (1.12)
  Week 3 | 4.61 (2.4) | 4.23 (1.85)
  Week 4 | 4.05 (2.3) | 3.98 (2.17)
  Week 5 | 3.84 (1.95) | 4.29 (1.99)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model includes random intercepts; beta estimate = 0.364, Standard Error of Mean 0.133 — Estimation parameter is beta estimate for group by visit interaction term

5. Primary Outcome: Ratings of Withdrawal Symptoms During Smoking Abstinence, as Measured by the Minnesota Tobacco Withdrawal Scale (MNWS)
Description: as for outcome 3
Time Frame: Baseline (pre-intervention) abstinence session (i.e., prior to week 1), follow-up abstinence session (immediately after final week of cigarette use; i.e., week 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 (pre-intervention) abstinence session | 13.2 (5.8) | 14.4 (4.56)
  Week 5 (post-intervention) abstinence session | 8.63 (5.93) | 11.6 (4.66)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.325, Mixed Models Analysis — Group is entered as a between-subjects factor and Visit is included as a repeated factor with 2 levels (pre- vs post-intervention). Baseline pain and FTCD scores, assessed at screening, are included along with sex as covariates; Model includes random intercepts; beta estimate = 1.78, Standard Error of Mean 1.78 — Estimation parameter is beta estimate for group by visit interaction term

6. Primary Outcome: Pain Intensity During Smoking Abstinence as Measured by the Past 24-hour Version of the Brief Pain Inventory (BPI)
Description: as for outcome 4
Time Frame: Baseline (pre-intervention) abstinence session (i.e., before week 1), follow-up abstinence session (immediately after final week of cigarette use; i.e., week 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 (pre-intervention) abstinence session | 4.53 (2.06) | 3.83 (1.78)
  Week 5 (post-intervention) abstinence session | 3.51 (2.26) | 2.85 (1.64)

7. Other Pre Specified Outcome: Changes in Smoking to Cope With Pain as Measured by the Pain and Smoking Inventory (PSI)
Description: The PSI is a 9-item measure of pain as a motivator to smoke, smoking to cope with pain, and pain as a barrier to smoking cessation, with responses indicated on a 7-point likert scale ranging from 0 (not true at all) to 6 (extremely true). Scores are averaged and the total score ranges from 0-6, with higher scores indicating that pain is a greater motivator to smoke.
Time Frame: Weekly visits 1, 3, and 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 | 2.87 (1.79) | 2.29 (1.16)
  Week 3 | 2.61 (1.77) | 2.52 (1.46)
  Week 5 | 2.13 (1.86) | 2.44 (1.33)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.035, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model includes random intercepts; beta estimate = 0.222, Standard Error of Mean 0.104 — Estimation parameter is beta estimate for group by visit interaction term

8. Other Pre Specified Outcome: Changes in Motivation to Quit Smoking as Measured by the Contemplation Ladder
Description: The contemplation ladder is a single-item measure of a person's current thoughts about quitting smoking, ranging from 0 (I have no thought of quitting) to 10 (I am doing something to try to quit)
Time Frame: Weekly visits 1, 3, and 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 | 5 (3.06) | 3.88 (2.55)
  Week 3 | 5.26 (2.75) | 5.31 (2.57)
  Week 5 | 5.95 (3.06) | 5.63 (3.18)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.27, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model includes random intercepts; beta estimate = 0.201, Standard Error of Mean 0.181 — Estimation parameter is beta estimate for group by visit interaction term

9. Other Pre Specified Outcome: Changes in Smoking Abstinence Self-efficacy as Measured by the Smoking Self-Efficacy Questionnaire (SEQ-12)
Description: The SEQ-12 is a 12-item measure yielding scores for self-efficacy when faced with both external (situational) or internal (e.g., affective) stimuli. Responses on each item range from 1 to 5, with higher scores indicating greater confidence in abstaining from smoking. Total score ranges from 12 to 60.
Time Frame: Weekly visits 1, 3, and 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 | 24.11 (6.88) | 27.44 (11.12)
  Week 3 | 29.68 (11.72) | 31 (8.92)
  Week 5 | 27.21 (8.64) | 25.63 (6.51)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.24, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model includes random intercepts; beta estimate = -1.229, Standard Error of Mean 1.037 — Estimation parameter is beta estimate for group by visit interaction term

10. Other Pre Specified Outcome: Pain Intensity Ratings During Ecological Momentary Assessment
Description: Responses to the question "Right now, how intense is your pain?", rated on a 1 (not at all) to 9 (extremely) likert scale at multiple timepoints throughout the day over the course of a week. All responses recorded within a week (up to 35 per participant) were averaged to create a single value ranging from 1 to 9, with higher scores indicating more pain.
Time Frame: Baseline (pre-randomization; i.e., week 1) and the first and last weeks of study cigarette use (i.e., weeks 2 and 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
units on a scale
  Week 1 (Baseline) | 4.40 (1.88) | 3.23 (1.54)
  Week 2 | 4.23 (2.06) | 3.09 (1.55)
  Week 5 | 3.67 (2.10) | 3.05 (1.57)

11. Other Pre Specified Outcome: Smoking Urge Ratings During Ecological Momentary Assessment
Description: Responses to question "How strong is your current urge to smoke?", rated on a 1 (not strong at all) to 9 (extremely strong) likert scale, assessed at multiple timepoints each day. All responses recorded within a week (up to 35 per participant) were averaged to create a single value ranging from 1 to 9, with higher scores indicating greater smoking urge.
Time Frame: Baseline (pre-randomization; i.e., week 1) and the first and last weeks of study cigarette use (i.e., weeks 2 and 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
units on a scale
  Week 1 (Baseline) | 4.74 (2.47) | 3.78 (2.26)
  Week 2 | 4.43 (2.32) | 3.40 (2.09)
  Week 5 | 3.23 (2.33) | 3.98 (2.39)

12. Other Pre Specified Outcome: Negative Affect Ratings During Ecological Momentary Assessment
Description: Average of responses to 4 negative affect items (anxious, irritable, guilty sad) using the question prompt, "Right now, how much are you feeling...?", rated on a 1 (not at all) to 9 (extremely) likert scale, assessed at multiple times per day. All responses recorded within a week (up to 35 per participant) were averaged to create a single value ranging from 1 to 9, with higher scores indicating greater negative affect.
Time Frame: Baseline (pre-randomization; i.e., week 1), and the first and last weeks of study cigarette use (i.e., weeks 2 and 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
units on a scale
  Week 1 (Baseline) | 2.44 (1.21) | 1.89 (0.91)
  Week 2 | 2.98 (1.61) | 1.91 (1.13)
  Week 5 | 2.43 (1.60) | 2.05 (1.03)

13. Other Pre Specified Outcome: Intent to Smoke During Ecological Momentary Assessment
Description: Proportion of "yes" responses to question "Are you about to smoke a cigarette right now?", assessed multiple times during the day. Total "yes" responses were divided by total observations within each week to calculate proportion of responses.
Time Frame: Baseline (pre-randomization; i.e., week 1) and the first and last weeks of study cigarette use (i.e., weeks 2 and 5)
Measure: Mean (Standard Deviation); unit: proportion of responses
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
proportion of responses
  Week 1 (Baseline) | 0.35 (0.48) | 0.26 (0.44)
  Week 2 | 0.38 (0.49) | 0.30 (0.46)
  Week 5 | 0.21 (0.41) | 0.32 (0.47)

14. Post Hoc Outcome: Changes in Abstinence-induced Craving as Measured by the Questionnaire of Smoking Urges-Brief (QSU-Brief)
Description: The QSU-Brief is a 5-item measure of urge to smoke, with responses indicated on a 7-point likert scale ranging from 0 (strongly disagree) to 7 (strongly agree). Total scores range from 0 to 35, with higher scores indicating greater craving.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLNC Group | NNC Group
Number analyzed (Participants) | 19 | 16
score on a scale
  Week 1 (pre-intervention) abstinence session | 26.3 (5.75) | 26.7 (6.34)
  Week 5 (post-intervention) abstinence session | 16.7 (9.42) | 21.8 (7.57)
Statistical Analysis 1: Comparison: VLNC Group vs NNC Group; Test type: Superiority; p = 0.113, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; Model includes random intercepts; beta estimate = 4.69, Standard Error of Mean 2.88 — Estimation parameter is beta estimate for group by visit interaction term

ADVERSE EVENTS:
Time Frame: 5 weeks including 1 week pre-randomization (abstinence 1 to weekly visit 1) and 4 weeks of study cigarette use (weekly visit 1 abstinence 2)
Arm/Group | VLNC Group | NNC Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 12/19 | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VLNC Group (N=19) | NNC Group (N=16)
dental extraction (Surgical and medical procedures) | 1 | 0
depressive symptoms (Psychiatric disorders) | 1 | 0
nausea and dizziness (Gastrointestinal disorders) | 0 | 2
100% increase in cigarettes/day (Product Issues) | 0 | 1
Elevated blood pressure (Vascular disorders) | 3 | 3
Fall, hurt ribs (Injury, poisoning and procedural complications) | 0 | 1
dizziness and blurred vision (Nervous system disorders) | 0 | 1
pinched nerve in hand (Nervous system disorders) | 1 | 0
heartburn (Gastrointestinal disorders) | 1 | 0
irregular heartrate (Cardiac disorders) | 1 | 0
tingling in chest (Nervous system disorders) | 1 | 0
knee, joint, or shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 5
mild pain in sternum (Musculoskeletal and connective tissue disorders) | 0 | 1
sinus irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
viral infection (Infections and infestations) | 1 | 0
increased stress (Social circumstances) | 2 | 1
increased anxiety (Psychiatric disorders) | 2 | 3
increased irritability (Psychiatric disorders) | 1 | 0
increased back pain (Musculoskeletal and connective tissue disorders) | 5 | 6
thyroid flare-up (Endocrine disorders) | 0 | 1
abcess (Infections and infestations) | 1 | 1
blocked salivary duct (Gastrointestinal disorders) | 0 | 1
Grief/sadness (Social circumstances) | 0 | 2
narcolepsy diagnosis (Nervous system disorders) | 1 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
minor back injury (Injury, poisoning and procedural complications) | 1 | 0
cirrhosis diagnosis (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT05032755/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT05032755/ICF_000.pdf